CLINICAL TRIAL: NCT04052074
Title: Complementary Therapy in Home Palliative Care Patients and Their Caregivers. A Clinical Trial
Brief Title: Complementary Therapy in Home Palliative Care Patients and Their Caregivers
Acronym: COMTHECARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Andaluz Health Service (Other Government)
Collaborators: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Principal Investigator, Francisco Javier Navarro Moya, Nurse Degree, Andaluz Health Service
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AP-0157-2018
Record Dates: First submitted 2019-07-14; First posted 2019-08-09 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Music Therapy; Caregivers; Palliative Care
Keywords: Music Therapy; Palliative Care; Caregivers; Nurses; Quality of Life; Cost efficiency analysis
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention group. Music in palliative patient (Experimental): Listening to pre-recorded and selected music preferred by the patient, half an hour for 7 days.
  Interventions: Other: Music Therapy
- Palliative patient. (Sham Comparator): Basic therapeutic education repetition performed to all patients through earphones, half, an hour for 7 days.
  Interventions: Other: simulation with therapeutic education
- Carer music. (Experimental): Listening to pre-recorded and selected music preferred by the carer, half an hour for 7 days.
  Interventions: Other: Music Therapy
- Carer. (Sham Comparator): Basic therapeutic education repetition performed to all carer through earphones, half an hour for 7 days.
  Interventions: Other: simulation with therapeutic education

INTERVENTIONS:
Other: Music Therapy — We are aiming to use music therapy, with pre-recorded favoured music, as a complementary treatment in oncological patients in palliative care, as well as on the carer. It will be performed using mp3 players or mobile phones.
  Arms: Carer music.; Intervention group. Music in palliative patient
Other: simulation with therapeutic education — Basic therapeutic education repetition performed to all caregivers and oncological patients in palliative care, through earphones
  Arms: Carer.; Palliative patient.

SUMMARY:
Introduction:

There is an increase on cancer prevalence and, consequently, a higher number of people that require palliative care, making an influence on the family and the main carer.

Objectives:

* To evaluate the efficiency and cost-effectiveness of a music intervention program, applied as a complementary therapy, in oncological palliative care patients and carers at home, compared to current treatment.
* To assess if patients in the intervention group submit significant differences regarding: pain, anxiety, depression, modo, insomnia, and life quality.
* To assess if carers in the intervention group present significant differences regarding the Caregiver Burden Scale and life quality.
* To evaluate patients and carers satisfaction on the therapeutic intervention.
* To estimate the cost-effectiveness of the intervention.

Method:

Randomised, double-blind, multi-centre clinical trial in the field of primary health care, conducted in 5 clinical management units belonging to Málaga-Guadalhorce health district and performed in oncological palliative care patients and carers. Two samples of 40 palliative care patients and two samples of 41 carers. The intervention group will undergo a 7-days intervention with music sessions, the control group will be given seven sessions of retraining in therapeutical education. Objectives will be evaluated through the following tools: Edmonton Scale, Symptom Assessment System, EORTC QLQ-C30, Caregiver Burden Scale, Pittsburgh Sleep Quality Index, Accelerometer, Epworth Sleepiness Scale (ESS), The Quality of Life Family Version, Client Satisfaction Questionnaire and Economical valuation.

To assess the objectives evaluations will be performed through home visit, both pre-intervention and a week after the beginning of the intervention for both groups. A follow-up visit will be made a month after the intervention to regard some economical parameters.

Statistical analysis:

The basal values of both groups will be compared. These values will be compared before and after the intervention, in the control and intervention group through Student t-test for normal continuous variables, and through Wilcoxon t-test for paired data in not normal continuous variables. In addition to the bivariated analysis, a multiple lineal regression will be carried out. The economical valuation will be a cost-effectiveness analysis. For each group we will measure cost, incremental cost, AVAC effectiveness, incremental effectiveness, dominance and, in case there is none, the results will be expressed in terms of incremental cost-effectiveness. To assess the costs, direct sanitary costs and intervention related costs will be considered.

SPSS 23 will be the statistical software to use, along with Epidat 3.01. 95% confidence range will make p values under 0,05 (p<0.05) statistically significant.

DETAILED DESCRIPTION:
Background and status.

Cancer presents an enormous challenge to the world public health. Every year, 8 million people die because of the disease, meaning it´s one of the main causes of death in the world and the pathology changes the patient in all their levels: physical (appearance, treatment consequences), emotional (reactions variability, feelings, distress), cognitive (personality and character, ways of facing the problem and adaptability), social and spiritual. It produces suffering on an individual, familiar and social level.

An estimation of 50-60% of the people that perish in Spain, based on age and death causes, does so after the disease reaches an advanced stage, being terminal. Terminal patients require great amounts of nursing and health care, being these needs very heterogenic and implying both sanitary and social resources.

According to the Andalusian Plan for Palliative Care estimations, Andalusian population susceptible to receive palliative care stands between a minimum of 31.553 and a maximum of 62.887 inhabitants.

World Health Organization (WHO) defined palliative care as: 'An approach that improves the quality of life of patients and their families facing the problem associated with life-threatening illness, through the prevention and relief of suffering by means of early identification and impeccable assessment and treatment of pain and other problems, physical, psychosocial and spiritual'.

A revision carried out in 2011 by the World Federation of Music Therapy (WFMT) defined music therapy as 'The professional use of music and its elements as an intervention in medical, educational, and everyday environments with individuals, groups, families, or communities who seek to optimize their quality of life and improve their physical, social, communicative, emotional, intellectual, and spiritual health and wellbeing'.

Integrating music therapy into palliative care intervention could help patients and caregivers to deal with some of the physical, emotional, social and spiritual needs they face: making changes in pain and anxiety perception easier, improving the mood, relaxing, enabling better emotional expressions, connecting with spirituality and offering support during mourning.

To perform adequate care services at home, a main caregiver is needed to guarantee that patients have all their basic needs cover, follow the scheduled treatment for the symptoms, get continuous family and social support and attention, specially at the end. But the caregiver's health can be affected, specially if subjected to an overload of work or adaptation to rapid changes in the person taken care of, affecting its quality of life.

For the most optimal performance of the caregiver, it is needed that they are also recognised. A systematic review in 2008 showed a lack of evidence-based interventions that support attention given to the caregivers of cancer patients, encouraging nurses to keep researching and putting to test intervention that reduce the burden on caregivers. However, several interventions in the attention to caregivers of terminal or palliative care patients proves their efficacy. Regarding the use of music therapy to achieve an improvement on the caregiver wellbeing, very few studies can be found.

Bibliography offers more and more studies and systematic reviews regarding music therapy in the intervention of cancer patients under palliative care, where the main goal is the study of the music therapy as a complementary treatment and a no-pharmacological treatment of anxiety, depression, pain, quality of life and physiological symptoms, pointing to its efficacy.

Kordovan et al. (2016) performed a prospective review of viability, acceptance and possible beneficial effects of music therapy in hospitalised terminal cancer patients, and the authors summarised that music therapy, especially receptive methods, are feasible and well regarded among these patients. A controlled randomised trial performed with hospitalised palliative care patients revealed music therapy to be an effective treatment to promote relaxation and wellbeing for the patients. The music therapy didn't differ from the control treatment in terms of pain reduction, but it was significantly different in the fatigue aspect of quality of life scale , being considerably lower. Control treatment was verbal relaxation.

On economic aspects, Keenan A., Keithley JK. (2015) made an integrating review about music effect in adults' cancer pain, stating a limited evidence of music therapy in pain treatment. Integrative methods using music may represent an important intervention that nurses can suggest as an economical, non-toxic and easily available to potentially reduce cancer pain. Efficiency wise, several publications point to a reduction in expenses mainly due to a lower medication intake, and it may as well mean a reduced number of professional attention and hours dedicated to deal with the symptoms.

Another systematic review by Qi He Mable L., Drury VB., Hong PW. (2010) showed the development of two important finding: music therapy can and must be used in palliative environments to promote social interaction and communication with family, friends, other patients and health practitioners; and it may as well be used to provide support to patients' needs. Through music therapy, patients noticed an improvement on social interaction and communication with their surroundings and a better way to satisfy their physical, psychological and spiritual needs.

In a Cochrane review from Bradt et al. (2016), authors concluded that music intervention can bring positive results on anxiety, pain, mood and quality of life in cancer patients, but the results must be read with caution as the bias risk is high.

In a study carried out by Gallager et al. (2017), it was proposed to understand the insight of family members regarding music therapy undertaken by the palliative care patients. Out of 50 participants, 82% indicated an improvement for both the relative and the patient in stress management, mood and quality of life, the session being rated as extremely useful in the 80% of cases, and 100% of them recommended more sessions. Patients reported a statistically significant improve regarding pain, depression, distress and mood. The study concludes that palliative patients´ relatives inform of an improvement on both patients and relatives, but more research is needed to fully comprehend the beneficial effects on the family.

This study proposes using music therapy on both patients and caregivers, differing in the way of choosing the music. Whereas most studies in the bibliography resort to picking relaxing music among different categories, such as jazz, folk or country, we aim to ask the participants to choose the music the want to listen to. This study will consider that the same genre can vary in the options available for the patients, triggering different emotions in different people depending on personal experiences. Although people can distinguish between sad and cheerful tunes, most people have preferred music that cheer us up or saddens us and we use it to our convenience, so the study will focus on the music that makes each patient feel better, assuming than that is the key to achieve better results.

This clinical trial will consider all recommendations from the authors of the Cochrane 2016 review to avoid bias.

Despite the high potential benefit that it could be to optimise medication intake and reduce sanitary resources expenditure, the evidence on cost-effectiveness in music intervention is very limited, so this study will also try to determine the efficiency of the intervention. Economic evaluation methods will be applied, along with a helping tool to determine, through decisions taken, the optimal use of sanitary resources and allowing the gathering of feedback of the impact of the intervention for both the organisation and the social program.

General objective:

- To evaluate the efficacy and cost-effectiveness of a music intervention program applied as a complementary treatment on palliative care for oncological patients and caregiver in a domestic environment, compared to standard treatment.

Specific objectives:

* To assess if the oncological patients in palliative care included in the intervention group present significant differences with the control group regarding: pain, anxiety, depression, mood and insomnia.
* To evaluate if the oncological patients in palliative care included in the intervention group present significant differences with the control group in their quality of life.
* To assess if the caregivers of the intervention group patients present significant differences with those of the control group regarding the Caregiver Burden Scale and quality of life.
* To value caregivers and patients' satisfaction with the intervention.
* To estimate the sanitary cost associated to the music intervention program compared to traditional sanitary interventions.

Methodology:

Randomised, double-blind, multi-centre clinical trial in the field of primary health care, conducted in 5 clinical management units belonging to Málaga-Guadalhorce health district and performed in oncological palliative care patients included into the Assistance Procedure of Palliative Care in digital health history (DIRAYA) and their unofficial caregivers.

* Subjects acquisition will be performed randomly through a phone list obtained using the program Epidat 3.1, taking the required number of palliative care patients, contacting each of them and evaluating if inclusion criteria are met, offering the chance of taking part of the intervention and handing over the correspondent information document. In case the patient accepts, a consent form must be signed. In case the patient has an unofficial caregiver, they will be offered to take part in the study as well, giving them the information sheet and signing the consent form specific for the caregiver in case they accept.
* The randomisation mechanism that has been chosen is as follows: letters will be ready with 'you have been included in the intervention group' and 'you have been included in the control group' in a number that meet the requirements, they will be put into opaque envelopes, shuffled and numbered. Participants will be assigned a participation number and the researcher in charge of randomisation will pick and open the envelope assigned to the participant number. This system ensures the number is fixed for each group and prevents tampering.

The palliative care patient and the caregiver are offered to participate and, if both accept, they will be offered an envelope that will be valid for both, taking part into the study in the same group. If only one of the two accepts, they will be offered an envelope as well. Participants will be taken until the desired number of cases is reached.

Once the researcher in charge of randomisation knows which groups the patient and the caregiver belong to according to the envelope, they will be informed of the procedure they will undergo without knowing their belonging to either the control or the intervention group.

• Sample size: the most relevant variable to be considered is anxiety for palliative care patients. In Bradt et al. (2016) revision it was presented with a standard deviation of 1'8 in a similar sample using a scale with a wider range than the one used in this study. Previous bibliography shows significant differences after music intervention, with a specific estimation of difference in 7 (29% of standard deviation). A research using the Edmonton Scale (in oncological patients, treatments with ginseng) showed a value of 0-83 points with a standard deviation of 2.34 (35% of standard deviation). If we consider as clinically relevant a decrease of 2 points in the anxiety before-after, expecting a standard deviation of at most 2.5 in our population; with an alpha error of 0.05 and a beta of 0.10 2 samples of 33 subjects are needed, choosing the ration for the samples in 1:1. A 20% increase, making it 2 samples of 40 subjects, would be desirable to avoid patients loss/dropping the intervention.

According to Hanser et al. (2011), there is an increase in the caregivers´ satisfaction with the music therapy, with a standard deviation of 1.33 on relaxation, 1.87 on comfort, and 1.23 in happiness. If we take a 1-point increase in caregivers' happiness as relevant, 2 samples of 34 carers would be needed. A 20% increase, making it 2 samples of 41 subjects would be desirable to avoid subjects loss/dropping the intervention.

* Procedures by group

  * Control group: the regular treatment will be carried out according to the Andalusian Plan of Palliative Care of the Health Counsel, following the standards and recommendations from the Minister of Health and Social Policy Palliative Care Units. It will consist on a complete initial valuation of the palliative care patient and the caregiver using Virginia Henderson's 14 fundamental needs (Need Theory) and the subsequent treatment and follow-up care plan for problems and symptoms detected; a therapeutic education about eating and hydration, lessons about exercise and leisure, medication, effective communication, skin care, prevention and treatment of constipation, and sleep hygiene will be also carried out. These patients and caregivers will receive the basic therapeutic education in a mp3 player or mobile phone (audio document shared on Drive) to be repeated and listened to in daily sessions of 30 minutes for 7 days. This way, the patients won´t know the group they are included in, and the nurses managing and evaluation the patients will also be blind.
  * Intervention group: subjects will receive conventional health assistance, complemented by music therapy activity consisting in pre-recorded preferred music, for both patients and caregivers. Music will be chosen among the one that make each of the subjects feel good. It will be reproduced through an mp3 player or mobile phone (using the Premium Spotify program) in daily sessions of 30 minutes for 7 days.
* To evaluate the expected objectives, valuations by means of home visits will be made, both preintervention and a week after the start of the intervention, for both groups. A home visit will also be done after a month to assess economic parameters.
* The following valuation scales will be used: Edmonton Scale, Symptoms Assessment System, EORTC QLQ-C30, Caregiver Burden Scale, Pittsburgh Sleep Quality Index, Epworth Sleepiness Scale (ESS), The Quality of Life Family Version, Client Satisfaction Questionnaire, and Economic valuation.
* Statistical analysis: a descriptive study of the collected factors will be carried out by means of media and standard deviation for normal continuous variables; calculating confidence interval for punctual estimations; through median and interquartile range in not normal continuous variables; and frequencies and percentages in categoric variables. Adjustment to normality will be determined by the Shapiro-Wilk test. The basal values of both groups will be compared before and after the intervention, in the control and intervention group through Student t-test for normal continuous variables, and through Wilcoxon t-test for paired data in not normal continuous variables. In addition to the bivariated analysis, a multiple lineal regression will be carried out, where the dependant variables will be: pain, anxiety, depression, mood, insomnia and quality of life; the independent variables will include intervention, sociodemographic (sex, age, studies, civil status) and clinical (pathology, palliative care time) variables of the subjects. The economic valuation will be a cost-effectiveness analysis, following the recommendations proposed in the guide to evaluate economic performances in health technologies. For each group, we will measure the cost, incremental cost, AVAC effectiveness, incremental effectiveness, dominance and, in case there is no dominance, results will be showed as an incremental cost-effectiveness ratio. To assess the costs, direct sanitary costs and intervention related costs will be considered. Sanitary resources costs will be estimated using the public prices set by the SSPA58. The cost of direct resources used during the intervention will be estimated by means of their recommended retail price (RRP). To calculate the AVAC, the EuroQol-5D-5L Questionnaire will be used. Uncertainty variables analysis will be subject to univariant and polyvariant sensitivity analysis.

In the event of finding statistically significant data in normal variables, the confidence range will be calculated on 95%, allowing the estimation of values where the difference is found. SPSS will be the statistical software to use, along with Epidat 3.01. 95% confidence range will make p values under 0,05 (p<0.05) statistically significant.

• This study is in agreement with the current ethic recommendations:

* Principles of the Declaration of Helsinki (1975) reviewed in 2013 (AMM), ethical principles for researching in human, adopted by the 64th Genera Assembly, Fortaleza, Brazil, October 2013).
* All personal data and information obtained in this study are confidential and will be deal with in accordance to the EU regulation 2016/679 of the European Parliamentary Group and the Council on April 27th of 2016 for General Data Protection Regulation (GDPR).
* Law 41/2002 from November 14th, basic regulation law for patient´s autonomy, obligations and rights regarding information and clinical documentation. Participation will be voluntary, and a written consent form must be signed to be included in the study. Patients and caregivers will be treated with maximum respect, without economic, religious, ethnic or sexual orientation discrimination. All participants will be informed both oral and written about the content and characteristics of the study, remarking the voluntary character and the possibility of rejecting taking part in the study, or dropping from it in any moment if it is desired. All data obtained will be private and confidential, its use reserved only for the purposes of this study and being destroyed afterwards.

The investigation Project hast been accepted by the Ethic Committee for Provincial Research in Malaga. During the study, the Code of Good Scientific Practice will be upheld.

ELIGIBILITY:
Inclusion Criteria:

* Oncological patients in palliative care at their homes, older than 18 years old, and their formal caregiver, in case they have one.
* Patients who have given their consent to be included in the study.

Exclusion Criteria:

* Oncological patients in palliative care at their homes, with diseases in an advanced stage and a short life expectancy (last days).
* Oncological patients with late stages dementia or psychological pathologies, not being capable of taking conscious decisions.
* Oncological patients with hypoacusis or profound deafness, hindering the use of the mp3 player or mobile phone.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-09-20 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the change of symptoms (at the beginning and at 7 days) using The Edmonton Symptom Evaluation System (ESAS) | Preintervention/Postintervention (0 and 7 days)
  This scale evaluates the average intensity for several symptoms (pain, anxiety, depression, mood and insomnia) in a specific length of time (24 hours, 48 hours, a week) dependant on the patient's condition. The patient will choose the number that better adjust to the intensity of each symptom.
Evaluation of the change in health-related quality of life (at the beginning and at 7 days) through The EORTC. QLQ-30 (The Quality of Life of Cancer Patients).Version 3 | Preintervention/Postintervention ( 0 and 7 days)
  Questionnaire to assess the quality of life of cancer palliative care patients, constituted by 30 items. Items from 1 to 28 correspond to mixed categoric scales from 1 to 4 referring to functional status, physical and emotional symptoms, and the influence of these in the working, social and familial life of the patient. Items 29 and 30 are for the patient to evaluate its general health and quality of life with a 0 to 7 mark.
Evaluation of the change in the caregiver's effort index (at the beginning and at 7 days) through The Caregiver Strain Index Questionnaire (CSI) | Preintervention/Postintervention ( 0 and 7 days)
  Aimed to be answered by the caregiver of dependent people, containing 13 items with True/False answer. Every positive answer scores for 1. If the total is higher or equal to 7 it indicates a high level of strain. Being validated in Spanish, this is the scale used to evaluate the emotional and physical situation of the caregiver regarding their need to take care of a person in palliative care.
Client Satisfaction Questionnaire (CSQ-8) | Postintervention (7 days)
  8 questions answered through a Likert-type scale of 4 points and self-administered, with specific points to each item. The categories would be as follows: quality of the service, type of services, results and general satisfaction. It will include 3 open questions where the subjects answer what they liked most from the treatment, what they liked less, and what they would change. This tool has been proved to determine patient´s satisfaction with high reliability and coherence, being validated in the 8 items versions for Spanish speakers.
Evaluation of the change in the quality of self-perceived sleep (at the beginning and at 7 days) through The Pittsburgh Sleep Quality Index (PSQI) | Preintervention/Postintervention ( 0 and 7 days)
  Validated into Spanish. It values the sleep quality perceived by the subject. 7 different scores are obtained from the result, granting information for several components of the sleep quality: subjective quality, sleep latency, sleep duration, sleep efficiency, sleep perturbances (frequency of coughs, snores, heat, cold), sleeping pills intake, diurnal dysfunction (faculty to fall asleep through an activity because of tiredness). The sum of the scores in each component will be included into a Total Score (TS) from 0 to 21. According to Buysse and Cols, a TS of 5 will be the cutting point between a good and a bad sleep quality, less than 5 will show the presence of good sleep quality.
Evaluation of the change in total sleep time and rest time (nighttime sleep and daytime rest / naps) by accelerometer (at the beginning and at 7 days) | Preintervention/Postintervention (0 and 7 days)
  The accelerometer triaxial: (GeneActiv, Activinsight Ltd, Kimbolton, Cambs, UK, http://www.geneactiv.org/). The data processing is done with an open source package in R, GGIR version 1.5-12.
Evaluation of the change in sleep interruption (number of awakenings and wakefulness after the onset of sleep) by accelerometer (at the beginning and at 7 days) | Preintervention/Postintervention ( 0 and 7 days)
  The accelerometer triaxial: (GeneActiv, Activinsight Ltd, Kimbolton, Cambs, UK, http://www.geneactiv.org/). The data processing is done with an open source package in R, GGIR version 1.5-12.
Evaluation of the change in sleep efficiency (percentage of time in bed sleeping) (at the beginning and at 7 days) by accelerometer | Preintervention/Postintervention ( 0 and 7 days)
  The accelerometer triaxial: (GeneActiv, Activinsight Ltd, Kimbolton, Cambs, UK, http://www.geneactiv.org/). The data processing is done with an open source package in R, GGIR version 1.5-12.
Evaluation of the change in the levels of intensity of daily physical activity (at the beginning and at 7 days) by accelerometer | Preintervention/Postintervention ( 0 and 7 days)
  The accelerometer triaxial: (GeneActiv, Activinsight Ltd, Kimbolton, Cambs, UK, http://www.geneactiv.org/). The data processing is done with an open source package in R, GGIR version 1.5-12.
  When the EPOCHS (5-second sections) have been calculated, periods of different intensity levels are sought (both sedentary lifestyle maintained and intense activities maintained continuously for most of a period of time). With them, variables are created that indicate both sedentary lifestyle and physical activity.
Evaluation of the change in daytime sleepiness (at the beginning and at 7 days) through the Epworth Sleepiness Scale (ESS) | Preintervention/Postintervention ( 0 and 7 days)
  Self-administered scale to measure diurnal sleepiness with 8 questions, scoring from 0 to 3 for a maximum score of 24. This scale is validated in Spanish.
Evaluation of the change in the quality of life of the caregiver (at the beginning and at 7 days) through The Quality of Life Family Version (QOL). Dr | Preintervention/Postintervention ( 0 and 7 days)
  It is an instrument that measures the quality of life of a family member who is caring for a patient in chronic illness, validated to Spanish. It values physical and emotional aspects.
Evaluation of the consumption of health resources at the beginning, at 7 days and per month | Preintervention/ Postintervention/per month ( 0 and 7 days and one month after the intervention)
  To calculate the expenditure we will analyse the number of Primary Care consultations (family doctor and family nurse), number of home consultations (family doctor, family nurse and case management nurse), number of consultations to the Emergencies service in Primary Care, number of consultations to the hospital Emergencies, and number of hospital admissions (registering number of days). The time used by medical practitioners in phone calls will be also taken into account, from both the Palliative Care Unit and the case management nurse.
Medication consumption evaluation at the beginning, at 7 days and per month | Preintervention/ Postintervention/per month ( 0 and 7 days and one month after the intervention)
  We will value the medication intake related to analgesics, anxiolytics and sleeping pills.
Availability of payment | Postintervention (7 day)
  The contingent valuation method will be used to determine the readiness to pay. Patients
Sessions compliance. Assessment question | Postintervention (7 day)
  Real time dedicated to the activity, for both control and intervention group, will be asked to patients and caregivers during the home visit.

SECONDARY OUTCOMES:
Sociodemographic data from palliative care patients | Preintervention (0 day)
  Age, sex, civil status, education level, time in palliative care, and disease they receive the care for.
Sociodemographic data from caregivers | Preintervention (0 day)
  Age, sex, civil status, education level, out-of-home job, time dedicated to caring, help received for caring, total time taking care of someone, and relation to the person taken care of.

CONTACTS AND LOCATIONS:
Overall Officials: Inmaculada Valero Cantero, Nurse, Principal Investigator — Distrito Sanitario Málaga- Guadalhorce. Servicio Andaluz de Salud; Milagrosa Espinar Toledo, Nurse, Study Chair — Distrito Sanitario Málaga- Guadalhorce. Servicio Andaluz de Salud; Yolanda Carrión Velasco, Nurse, Study Chair — Distrito Sanitario Málaga- Guadalhorce. Servicio Andaluz de Salud; Pilar Castro López, Nurse, Study Chair — Distrito Sanitario Málaga- Guadalhorce. Servicio Andaluz de Salud; Milagros Reyes Sánchez, Nurse, Study Chair — Distrito Sanitario Málaga- Guadalhorce. Servicio Andaluz de Salud; María Angeles Vázquez Sánchez, Doctor, Study Chair — Universidad de Málaga; Nuria Garcia-Agua Soler, Doctor, Study Chair — Universidad de Málaga; Cristina Casals Vázquez, Doctor, Study Chair — University of Cadiz; Francisco Martínez Valero, Podólogo, Study Chair — Clinica de Podologia; Ernesto Suárez Cadenas, Doctor, Study Chair — Universidad de Granada; Librado Valverde, Nurse, Study Chair — Distrito Sanitario Málaga- Guadalhorce. Servicio Andaluz de Salud
Locations (1):
- Inmaculada Valero Cantero, Málaga, Spain

REFERENCES:
- [Result] Williams AL, McCorkle R. Cancer family caregivers during the palliative, hospice, and bereavement phases: a review of the descriptive psychosocial literature. Palliat Support Care. 2011 Sep;9(3):315-25. doi: 10.1017/S1478951511000265. PMID 21838952
- [Result] Kordovan S, Preissler P, Kamphausen A, Bokemeyer C, Oechsle K. Prospective Study on Music Therapy in Terminally Ill Cancer Patients during Specialized Inpatient Palliative Care. J Palliat Med. 2016 Apr;19(4):394-9. doi: 10.1089/jpm.2015.0384. Epub 2016 Feb 19. PMID 26894922
- [Result] Keenan A, Keithley JK. Integrative Review: Effects of Music on Cancer Pain in Adults. Oncol Nurs Forum. 2015 Nov;42(6):E368-75. doi: 10.1188/15.ONF.E368-E375. PMID 26488843
- [Result] Qi He Mabel L, Drury VB, Hong PW. The experience and expectations of terminally ill patients receiving music therapy in the palliative setting: a systematic review. JBI Libr Syst Rev. 2010;8(27):1088-1111. doi: 10.11124/01938924-201008270-00001. PMID 27820208
- [Result] Bradt J, Dileo C, Magill L, Teague A. Music interventions for improving psychological and physical outcomes in cancer patients. Cochrane Database Syst Rev. 2016 Aug 15;(8):CD006911. doi: 10.1002/14651858.CD006911.pub3. PMID 27524661
- [Result] Gallagher LM, Lagman R, Rybicki L. Outcomes of Music Therapy Interventions on Symptom Management in Palliative Medicine Patients. Am J Hosp Palliat Care. 2018 Feb;35(2):250-257. doi: 10.1177/1049909117696723. Epub 2017 Mar 9. PMID 28274132
- [Result] McConnell T, Scott D, Porter S. Music therapy for end-of-life care: An updated systematic review. Palliat Med. 2016 Oct;30(9):877-83. doi: 10.1177/0269216316635387. Epub 2016 Mar 4. PMID 26944533
- [Result] Porter S, McConnell T, Clarke M, Kirkwood J, Hughes N, Graham-Wisener L, Regan J, McKeown M, McGrillen K, Reid J. A critical realist evaluation of a music therapy intervention in palliative care. BMC Palliat Care. 2017 Dec 8;16(1):70. doi: 10.1186/s12904-017-0253-5. PMID 29221475
- [Result] Gallagher LM, Lagman R, Bates D, Edsall M, Eden P, Janaitis J, Rybicki L. Perceptions of family members of palliative medicine and hospice patients who experienced music therapy. Support Care Cancer. 2017 Jun;25(6):1769-1778. doi: 10.1007/s00520-017-3578-y. Epub 2017 Jan 19. PMID 28105524
- [Result] Northouse LL, Mood DW, Schafenacker A, Kalemkerian G, Zalupski M, LoRusso P, Hayes DF, Hussain M, Ruckdeschel J, Fendrick AM, Trask PC, Ronis DL, Kershaw T. Randomized clinical trial of a brief and extensive dyadic intervention for advanced cancer patients and their family caregivers. Psychooncology. 2013 Mar;22(3):555-63. doi: 10.1002/pon.3036. Epub 2012 Jan 31. PMID 22290823
- [Result] Sales CA, da Silva VA, Pilger C, Marcon SS. [Music in human terminality: the family members' conceptions]. Rev Esc Enferm USP. 2011 Mar;45(1):138-45. doi: 10.1590/s0080-62342011000100019. Portuguese. PMID 21445500
- [Result] Ullrich A, Ascherfeld L, Marx G, Bokemeyer C, Bergelt C, Oechsle K. Quality of life, psychological burden, needs, and satisfaction during specialized inpatient palliative care in family caregivers of advanced cancer patients. BMC Palliat Care. 2017 May 10;16(1):31. doi: 10.1186/s12904-017-0206-z. PMID 28486962
- [Derived] Valero-Cantero I, Casals C, Espinar-Toledo M, Baron-Lopez FJ, Martinez-Valero FJ, Garcia-Agua Soler N, Vazquez-Sanchez MA. Effect of Self-Chosen Music in Alleviating the Burden on Family Caregivers of Patients with Advanced Cancer: A Randomised Controlled Trial. Int J Environ Res Public Health. 2023 Mar 6;20(5):4662. doi: 10.3390/ijerph20054662. PMID 36901671
- [Derived] Valero-Cantero I, Martinez-Valero FJ, Espinar-Toledo M, Casals C, Baron-Lopez FJ, Vazquez-Sanchez MA. Complementary music therapy for cancer patients in at-home palliative care and their caregivers: protocol for a multicentre randomised controlled trial. BMC Palliat Care. 2020 May 2;19(1):61. doi: 10.1186/s12904-020-00570-9. PMID 32359361
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Cancer+family+caregivers+during+the+palliative%2C+hospice%2C+and+bereavement+phases%3A+a+review+of+the+descriptive+psychosocial+literature.+Palliat+Support+Care.
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/26894922
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Integrative+Review%3A+Effects+of+Music+on+Cancer+Pain+in+Adults
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/27820208
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/27524661
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/28274132
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/26944533
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=A+critical+realist+evaluation+of+a+music+therapy+intervention+in+palliative+care
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/28105524
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Randomized+clinical+trial+of+a+brief+and+extensive+dyadic+intervention+for+advanced+cancer+patients+and+their+family+caregivers.
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Music+in+human+terminality%3A+the+family+members%27+conceptions.
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Quality+of+life%2C+psychological+burden%2C+needs%2C+and+satisfaction+during+specialized+inpatient+palliative+care+in+family+caregivers+of+advanced+cancer+patients